CLINICAL TRIAL: NCT00953849
Title: Vitamin D Plus Celecoxib Therapy to Stimulate Intratumoral Immune Reactivity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLIN-003-09S
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Mouth Neoplasms
Keywords: Calcitriol; Celecoxib; Immunotherapy
MeSH Terms: conditions — Mouth Neoplasms | interventions — Celecoxib; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: Celecoxib (Experimental): Celecoxib treatment prior to surgery
  Interventions: Drug: Celecoxib
- Arm 2: Calcitriol (Experimental): Treatment with Calcitriol prior to surgery
  Interventions: Drug: Calcitriol
- Arm 3: Celecoxib plus Calcitriol (Experimental): Treatment with Celecoxib plus Calcitriol prior to surgery.
  Interventions: Drug: Celecoxib plus Calcitriol
- Arm 4: No Treatment (No Intervention): no treatment prior to surgery

INTERVENTIONS:
Drug: Celecoxib — Celecoxib (400 mg twice daily)
  Other Names: Celebrex
  Arms: Arm 1: Celecoxib
Drug: Calcitriol — 3 week pre-surgical enteral treatment of Calcitriol (1,25-dihydroxyvitamin D3) (3 cycles of 4 microg Calcitriol 3 for each of 3 sequential days followed by 4 days of no treatment)
  Other Names: 1,25-dihydroxyvitamin D3
  Arms: Arm 2: Calcitriol
Drug: Celecoxib plus Calcitriol — 3 week pre-surgical enteral treatment of Calcitriol (1,25-dihydroxyvitamin D3) (3 cycles of 4 microg Calcitriol for each of 3 sequential days followed by 4 days of no treatment) plus Celecoxib (400 mg twice daily)
  Other Names: 1,25-dihydroxyvitamin D3
  Arms: Arm 3: Celecoxib plus Calcitriol

SUMMARY:
The poor survival of Veterans with oral cancer underscores the significance of identifying new treatment approaches. The proposed studies will test a new 2 pronged immunotherapeutic approach for oral cancer patients which lessen the immune inhibitory environment while maturing cells that can stimulate T cell reactivity against oral cancer cells.

DETAILED DESCRIPTION:
The hypothesis of this study is beneficial T cell reactivity in oral squamous cell carcinoma (OSCC) tumors can be synergistically stimulated by blocking suppressor endothelial cells and their induction of other inhibitory cell populations while also maturing immune inhibitory CD34+ cells into antigen-presenting dendritic cells.

To test this hypothesis, newly diagnosed OSCC patients will be administered the cyclooxigenase 2 inhibitor celecoxib and/or Calcitriol for the 3 week duration between cancer diagnosis and surgical treatment. The following aims will test the immunological and clinical effectiveness of the combination treatment:

* 1. To block the suppressive activity of endothelial cells and increase the levels of dendritic that are stimulatory to T cell reactivity, thereby synergistically increasing intratumoral T cell reactivity. These functional immune analyses will use OSCC tissues removed from untreated patients or patients treated with celecoxib and/or Calcitriol.
* 2. To reduce development of OSCC recurrences by synergistically stimulating intratumoral T cell reactivity with celecoxib to block suppressor endothelial cell activity and Calcitriol to mature CD34+ suppressor cells into T cell stimulatory dendritic cells.

ELIGIBILITY:
Inclusion Criteria:

* locoregional OSCC (T stage II-IV) of the oral cavity, oropharynx, larynx, or hypopharynx without evidence of distant metastases
* greater than or equal to 18 years of age
* the OSCC treatment plan includes surgical resection
* performance status of 0 or 1
* recovered from any prior surgery
* must be willing to use appropriate contraception if of child-bearing potential
* give signed informed consent prior to the initiation of therapy

Exclusion Criteria:

* prior immunotherapy
* chemotherapy or radiation therapy within three weeks
* concurrent NSAID treatments while undergoing treatment
* women pregnant or lactating
* HIV positive
* have an active infection requiring antibiotic therapy, or concomitant malignancies
* history of idiopathic urinary calcium stone disease, chronic hypercalcemia, or gastrointestinal malabsorptive conditions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Rita I Young, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication of deidentified results.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Celecoxib: Treatment with Celecoxib
- Arm 2: Calcitriol: Treatment with Calcitriol
- Arm 3: Celecoxib Plus Calcitriol: Treatment with Celecoxib + Calcitriol
Period: Overall Study
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment
Started | 6 | 6 | 4 | 5
Completed | 6 | 6 | 4 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Celecoxib: Celecoxib:
  Celecoxib (400 mg twice daily) oral cancer patients receiving new immunotherapy prior to surgery
- Arm 2: Calcitriol: Calcitriol Calcitriol (1,25-dihydroxyvitamin D3): 3 week pre-surgical enteral treatment of Calcitriol (3 cycles of 4 microg Calcitriol for each of 3 sequential days followed by 4 days of no treatment)
- Arm 3: Celecoxib Plus Calcitriol: Celecoxib + Calcitriol 3 week pre-surgical enteral treatment of Calcitriol (3 cycles of 4 microg 1,25-dihydroxyvitamin D3) for each of 3 sequential days followed by 4 days of no treatment) plus Celecoxib (400 mg twice daily)
- Arm 4: No Treatment: oral cancer patients receiving no immunotherapy prior to surgery
- Total: Total of all reporting groups
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment | Total
Number analyzed (Participants) | 6 | 6 | 4 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 3 | 4 | 15
  >=65 years | 2 | 2 | 1 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 0 | 4
  Male | 6 | 3 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in IL-2 Levels
Description: Change in IL-2 stimulatory cytokine levels within tumor tissue.
Time Frame: baseline and 3 weeks
Population: Patients with head and neck squamous cell carcinoma.
Measure: Mean (Standard Error); unit: pg/100 gm protein
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment
Number analyzed (Participants) | 6 | 6 | 4 | 5
pg/100 gm protein | 1.8 (0.3) | 4.0 (0.4) | 7.9 (1.2) | 2.1 (0.2)
Statistical Analysis 1: Comparison: Arm 1: Celecoxib vs Arm 2: Calcitriol vs Arm 3: Celecoxib Plus Calcitriol vs Arm 4: No Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; A Student's t test was performed to determine significance of differences between each of two groups

2. Primary Outcome: Change in IFN-gamma Levels
Description: Change in IFN-gamma stimulatory cytokine levels within tumor tissue.
Time Frame: baseline and 3 weeks
Population: Patients with head and neck squamous cell carcinoma.
Measure: Mean (Standard Error); unit: pg/100 gm protein
Groups:
- Arm 1: Celecoxib: oral cancer patients receiving new immunotherapy prior to surgery
  1,25-dihydroxyvitamin D3: 3 week pre-surgical enteral treatment of 1,25(OH)2D3 (3 cycles of 4 microg 1,25(OH)2D3 for each of 3 sequential days followed by 4 days of no treatment)
- Arm 2: Calcitriol: oral cancer patients receiving new immunotherapy prior to surgery
  celecoxib: celecoxib (400 mg twice daily)
- Arm 3: Celecoxib Plus Calcitriol: oral cancer patients receiving new immunotherapy prior to surgery
  1,25-dihydroxyvitamin D3 + celecoxib: 3 week pre-surgical enteral treatment of 1,25(OH)2D3 (3 cycles of 4 microg 1,25(OH)2D3 for each of 3 sequential days followed by 4 days of no treatment) plus celecoxib (400 mg twice daily)
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment
Number analyzed (Participants) | 6 | 6 | 4 | 5
pg/100 gm protein | 1.9 (0.6) | 2.8 (1.1) | 6.3 (2.2) | 2.0 (0.3)
Statistical Analysis 1: Comparison: Arm 1: Celecoxib vs Arm 2: Calcitriol vs Arm 3: Celecoxib Plus Calcitriol vs Arm 4: No Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; A Student's t test was performed to determine significance of differences between each of two groups

3. Primary Outcome: Change in GM-CSF
Description: Change in GM-CSF stimulatory cytokine levels within tumor tissue.
Time Frame: baseline and 3 weeks
Population: Patients with head and neck squamous cell carcinoma.
Measure: Mean (Standard Error); unit: pg/100 gm protein
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment
Number analyzed (Participants) | 6 | 6 | 4 | 5
pg/100 gm protein | 3.8 (1.4) | 8.1 (1.9) | 14.3 (3.4) | 3.2 (0.9)
Statistical Analysis 1: Comparison: Arm 1: Celecoxib vs Arm 2: Calcitriol vs Arm 3: Celecoxib Plus Calcitriol vs Arm 4: No Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; A Student's t test was performed to determine significance of differences between each of two groups

4. Primary Outcome: Change in IL-6 Levels.
Description: Change in levels of immune inhibitory/inflammatory mediator IL-6 in tumor tissue.
Time Frame: baseline and 3 weeks
Population: Patients with head and neck squamous cell carcinoma.
Measure: Mean (Standard Error); unit: pg/100 gm protein
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment
Number analyzed (Participants) | 6 | 6 | 4 | 5
pg/100 gm protein | 39 (18) | 46 (21) | 29 (8) | 132 (46)
Statistical Analysis 1: Comparison: Arm 1: Celecoxib vs Arm 2: Calcitriol vs Arm 3: Celecoxib Plus Calcitriol vs Arm 4: No Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; A Student's t test was performed to determine significance of differences between each of two groups

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Arm 1: Celecoxib: oral cancer patients receiving Celecoxib prior to surgery
- Arm 2: Calcitriol: oral cancer patients receiving Calcitriol prior to surgery
- Arm 3: Celecoxib Plus Calcitriol: oral cancer patients receiving Celecoxib + Calcitriol prior to surgery
- Arm 4: No Treatment: oral cancer patients receiving no treatment prior to surgery
Arm/Group | Arm 1: Celecoxib | Arm 2: Calcitriol | Arm 3: Celecoxib Plus Calcitriol | Arm 4: No Treatment
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Difficulty in recruiting subjects that are eligible for the combination Celecoxib + Calcitriol treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes